CLINICAL TRIAL: NCT04060160
Title: Acne Detection Software (AcneDect); AcneDect: a Software to Detect Acne Lesions
Brief Title: Acne Detection Software (AcneDect)
Acronym: AcneDect
Status: Terminated | Type: Observational
Why Stopped: After careful consideration and review of the data, the study team has determined that it is in the best interest of all parties involved to conclude the study at this juncture.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00702; sp19Navarini
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Acne Lesions; Acne Vulgaris
Keywords: machine learning; self-learning software; image-detecting software
MeSH Terms: conditions — Acne Vulgaris | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self- learning software that can detect acne lesions — Self- learning software that can detect acne lesions from patients who take a picture of their face every single day for 3 months with a secure mobile phone.
Other: Patient reported outcomes — Collection of patient reported outcomes and clinical data via a mobile electronic case report form

SUMMARY:
This study is to create a self-learning software that can detect acne lesions. Patients take a picture of their face every single day for 3 months with a secure mobile phone and fill out a pre-designed questionnaire. After 3 months, the mobile will be collected back and the pictures will be evaluated by 3 dermatologists. The software is able to learn from the dermatologists' evaluation and -using machine learning- a mechanism that should be able to automatically detect acne to some extent will be established.

ELIGIBILITY:
Inclusion Criteria:

* Acne vulgaris

Exclusion Criteria:

* Refusal to participate

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients within the consultation service of Dermatologische Klinik, Universitätsspital Basel, that meet the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Pictures to train the AcneDect software | every single day from baseline for 3 months
  Collection of pictures to train the AcneDect software to detect change in acne lesions

SECONDARY OUTCOMES:
AcneDect questionnaire regarding acne burden (Visual Analogue Scale (VAS) scale ranging from "Not bad at all" to "Very bad") | every single day from baseline for 3 months
  Collection of patient reported outcomes via a mobile electronic case report form

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A. Navarini, Prof. Dr. MD, Principal Investigator — Dermatologische Klinik; Universitätshospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland